CLINICAL TRIAL: NCT04427761
Title: Health-Illness Transition Experiences Among Patients With Pancreatic Cancer
Brief Title: A Study of the Life Changes Experienced by Patients With Pancreatic Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Hunter College School of Nursing (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20-038
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
Keywords: Quality of Life; Health-Illness Transition; 20-038
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pancreatic cancer health-illness transition: In this prospective longitudinal correlational study, a convenience sample of patients with pancreatic cancer receiving chemotherapy will be asked to report on their health-illness transition experiences and their level of distress.
  Interventions: Behavioral: Measurement of Transitions in Cancer Scale (MOT-CA) Survey; Behavioral: Distress Thermometer Survey

INTERVENTIONS:
Behavioral: Measurement of Transitions in Cancer Scale (MOT-CA) Survey — These surveys will take 5-10 minutes to complete at two time-points, T0 (baseline) and T1 (four to six weeks after baseline visit) The patient will again complete the DT and MOT-CA at a chemotherapy treatment or clinic visit, if possible, or via a telephone call with the principal investigator in the event that there are no in-person visits scheduled (Time 1).
Behavioral: Distress Thermometer Survey — These surveys will take 5-10 minutes to complete at two time-points, T0 (baseline) and T1 (four to six weeks after baseline visit).The patient will again complete the DT and MOT-CA at a chemotherapy treatment or clinic visit, if possible, or via a telephone call with the principal investigator in the event that there are no in-person visits scheduled (Time 1).

SUMMARY:
The purpose of this study is to better understand what types of transitions people with pancreatic cancer face when they receive chemotherapy. Again, this study defines transition as a change in a life situation or a status that causes a change in a person's identity, role, behavior, or personal relationships. Examples of transitions include changes in sleeping habits, anxiety, employment, relationship with a higher power, and treatment goals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18 years of age and older
* primary language listed as English in electronic medical record
* biopsy proven diagnosis of pancreatic cancer
* within three months after initiating a chemotherapy regimen at the Rockefeller Outpatient Pavilion at MSKCC (patient may have previously received chemotherapy at an outside institution or may have received previous chemotherapy regimens at MSKCC).

Exclusion Criteria:

* previous history of cancer within the past five years, except for non-melanoma skin cancer, ductal carcinoma in situ breast cancer, and thyroid cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Extent of the change experienced by patients with pancreatic cancer | 4 to 6 weeks after baseline
  Descriptive statistics will be calculated at both time points using (part A on the MOT-CA) for each of the seven transition domains (physical, emotional, social, spiritual, cancer status, treatment, and approach) at both time points (Time 0 and Time 1).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Goldberg, RN, MSN, AGPCNP-BC, ACHPN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm